CLINICAL TRIAL: NCT05423262
Title: A Phase I/II Study of TRK-950 in Patients With Advanced Solid Tumors
Brief Title: A Study of TRK-950 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 950P1V03
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor; Melanoma
Keywords: Nivolumab-eligible solid tumor; Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 : TRK-950 (Experimental): * Solid Tumor
  * TRK-950 will be administered intravenously on days 1, 8, 15, and 22 of a 28-day cycle. Two dose levels will be explored during this Arm.
  Interventions: Biological: TRK-950
- Part 2 Cohort 1: TRK-950+Nivolumab (Experimental): * Nivolumab-eligible solid tumor
  * Nivolumab will be administered intravenously on days 1 and 15 of a 28-day cycle. TRK-950 will be administered as an intravenously infusion on days 1, 8, 15 and 22. After the administration of Nivolumab on days 1 and 15, TRK-950 will be administered as an intravenously infusion.
  Interventions: Biological: TRK-950; Drug: Nivolumab
- Part 2 Cohort 2: TRK-950+Nivolumab (Experimental): * Nivolumab-eligible solid tumor
  * Nivolumab will be administered intravenously on days 1 and 15 of a 28-day cycle. TRK-950 will be administered as an intravenously infusion on days 1 and 15. After the administration of Nivolumab on days 1 and 15, TRK-950 will be administered as an intravenously infusion.
  Interventions: Biological: TRK-950; Drug: Nivolumab
- Part 3: TRK-950 (Experimental): * Melanoma
  * TRK-950 will be administered intravenously on days 1, 8, 15, and 22 of a 28-day cycle.
  Interventions: Biological: TRK-950

INTERVENTIONS:
Biological: TRK-950 — 5 or 10 mg/kg administered intravenously over 60 minutes (weekly)
  Arms: Part 1 : TRK-950
Biological: TRK-950 — 10 mg/kg administered intravenously over 60 minutes (weekly)
  Arms: Part 2 Cohort 1: TRK-950+Nivolumab
Biological: TRK-950 — 20 mg/kg administered intravenously over 60 minutes (bi-weekly)
  Arms: Part 2 Cohort 2: TRK-950+Nivolumab
Drug: Nivolumab — 240 mg administered intravenously over 30 minutes (bi-weekly)
  Arms: Part 2 Cohort 1: TRK-950+Nivolumab; Part 2 Cohort 2: TRK-950+Nivolumab
Biological: TRK-950 — 10 mg/kg administered Intravenously over 60 minutes (weekly)
  Arms: Part 3: TRK-950

SUMMARY:
Part 1

• To determine the safety and tolerability of TRK-950 in patients with advanced solid tumors

Part 2

• To determine the safety and tolerability of TRK-950 in combination with nivolumab(NIVO) in patients with advanced solid tumors eligible for NIVO therapy

Part 3

• To determine the efficacy of TRK-950 in patients with advanced/recurrent unresectable melanoma, who received prior chemotherapy with dacarbazine(DTIC) and for whom no standard therapy exists

DETAILED DESCRIPTION:
This is an open-label phase I/II study and consists of three parts. In Part 1, patients with histologically and cytologically confirmed locally advanced or metastatic solid tumors who have been refractory or intolerant to standard therapies or for whom no standard therapy exists will receive two dose level of TRK-950. In Part 2, patients with histologically and cytologically confirmed locally advanced or metastatic solid tumors who are eligible for standard therapy with NIVO 240 mg alone administered at 2-week intervals will receive two dose level of TRK-950 in combination with Nivolumab. In Part 3, patients with histologically confirmed locally advanced unresectable or metastatic melanoma (excluding uveal melanoma), who received prior chemotherapy with DTIC and for whom no standard therapy exists will receive one dose level of TRK-950. The objectives of this study are to determine the safety, tolerability, pharmacokinetic (PK) profile and the incidence of the development of anti-drug antibodies (ADA) and neutralizing antibodies (NAb) against TRK-950.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Patients with histologically and cytologically confirmed locally advanced or metastatic solid tumors who have been refractory or intolerant to standard therapies or for whom no standard therapy exists. Part 2: Patients with histologically and cytologically confirmed locally advanced or metastatic solid tumors who are eligible for standard therapy with NIVO 240 mg alone administered at 2-week intervals.
* Part 3: Patients with histologically confirmed locally advanced unresectable or metastatic melanoma (excluding uveal melanoma), who received prior chemotherapy with DTIC and for whom no standard therapy exists
* Patients with life expectancy of at least 3 months after the start of study drug administration
* Patients aged >=18 years at the time of consent
* Patients who are able to provide written consent in person to be a subject of this study
* A negative pregnancy test before enrollment (if female of childbearing potential)

Exclusion Criteria:

* Patients with active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy
* Pregnant women (including those who are considered possibly pregnant based on history taking, etc. by physician) or breastfeeding women (interrupting breastfeeding to enroll is also not allowed)
* Patients who are unwilling or unable to comply with the protocol specified procedures
* Patients who are positive for human immunodeficiency virus (HIV) antibody
* Patients who meet any of the following conditions on hepatitis B virus (HBV) and hepatitis C virus (HCV) testing

  * Patients who are positive for hepatitis B surface antigen (HBsAg)
  * Patients who are positive for HCV RNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) (Part 1 and 2) | Up to Day 28
  Number of participants with DLTs will be determined.
Number of participants with adverse events (AEs) (Part 1 and 2) | through study completion, an average of 1 year
  Number of participants with AEs will be assessed.
Number of participants with adverse events of special interest (AESIs) (Part 1 and 2) | through study completion, an average of 1 year
  Number of participants with AESIs will be assessed.
Number of participants with serious adverse events (SAEs) (Part 1 and 2) | through study completion, an average of 1 year
  Number of participants with SAEs will be assessed.
Objective response rate (ORR) (Part 3) | Up to approximately 12 months
  Objective response rate (ORR) is defined as the percentage of patients who achieved either complete response (CR) or partial response (PR) as assessed by independent central review (ICR) per RECIST Version 1.1.

SECONDARY OUTCOMES:
Area under the concentration curve (AUC) of TRK-950 (Part 1 and 2) | through study completion, an average of 1 year
Maximum plasma concentration (Cmax) of TRK-950 (Part 1 and 2) | through study completion, an average of 1 year
Time to maximum plasma concentration (Tmax) of TRK-950 (Part 1 and 2) | through study completion, an average of 1 year
Terminal elimination half life (t1/2) of TRK-950 (Part 1 and 2) | through study completion, an average of 1 year
Total body clearance (CL) of TRK-950 (Part 1 and 2) | through study completion, an average of 1 year
Apparent volume of distribution (Vd) of TRK-950 (Part 1 and 2) | through study completion, an average of 1 year
Area under the concentration curve (AUC) of Nivolumab (Part 2 only) | through study completion, an average of 1 year
Overall survival (OS) (Part 3) | Up to approximately 12 months
  Overall survival (OS) is defined as time from the first date of TRK-950 administration until the date of death due to any cause.
Progression-free survival (PFS) (Part 3) | Up to approximately 12 months
  Progression-free survival (PFS) is defined as time from the first date of TRK-950 administration until progression per RECIST Version 1.1, or death due to any cause.
Best overall response (BOR) (Part 3) | Up to approximately 12 months
  Best overall response (BOR) is defined as the best response among all responses at each time point from the first date of TRK-950 administration until progression per RECIST Version 1.1.
Disease control rate (DCR) (Part 3) | Up to approximately 12 months
  Disease control rate (DCR) is defined as the percentage of patients with BOR of CR or PR or stable disease (SD) per RECIST Version 1.1.
Duration of response (DOR) (Part 3) | Up to approximately 12 months
  Duration of response (DOR) is defined as the duration between the date of first documented response (CR or PR) and the date of progression per RECIST Version 1.1, or death due to any cause.
Tumor change rate (Part 3) | Up to approximately 12 months
  Tumor change rate is defined as the percentage change in the sum of the longest diameters of target lesions, as assessed per RECIST Version 1.1, compared to baseline obtained at screening.

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Shinshu University Hospital, Matsumoto, Nagano
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - National Cancer Center Hospital, Chuo Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okano F, Saito T, Minamida Y, Kobayashi S, Ido T, Miyauchi Y, Wasai U, Akazawa D, Kume M, Ishibashi M, Jiang K, Aicher A, Heeschen C, Yonehara T. Identification of Membrane-expressed CAPRIN-1 as a Novel and Universal Cancer Target, and Generation of a Therapeutic Anti-CAPRIN-1 Antibody TRK-950. Cancer Res Commun. 2023 Apr 18;3(4):640-658. doi: 10.1158/2767-9764.CRC-22-0310. eCollection 2023 Apr. PMID 37082579